CLINICAL TRIAL: NCT02062632
Title: A Pilot, Double-Blind, Randomized, Two-Arm Crossover Study of Doxepin Versus Placebo for Esophagitis-Induced Pain in Patients Receiving Radiotherapy to the Thorax With or Without Chemotherapy
Brief Title: Doxepin Hydrochloride in Treating Esophageal Pain in Patients With Thoracic Cancer Receiving Radiation Therapy to the Thorax With or Without Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC13C1; NCI-2014-00253 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC13C1 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2018-11

CONDITIONS: Esophageal Carcinoma; Hypopharyngeal Carcinoma; Laryngeal Carcinoma; Lymphoma; Mesothelioma; Metastatic Malignant Neoplasm in the Lung; Metastatic Malignant Neoplasm in the Pleura; Metastatic Malignant Neoplasm in the Spinal Cord; Non-Small Cell Lung Carcinoma; Sarcoma; Small Cell Lung Carcinoma; Thymic Carcinoma; Thymoma; Thyroid Gland Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Lymphoma; Mesothelioma; Carcinoma, Non-Small-Cell Lung; Sarcoma; Small Cell Lung Carcinoma; Thymoma; Thyroid Neoplasms | interventions — Doxepin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (doxepin hydrochloride) (Experimental): Patients receive doxepin hydrochloride oral solution (swish, gargle for 30 seconds, and slowly swallow) on day 1. Patients then crossover to Arm II on day 3.
  Interventions: Drug: Doxepin Hydrochloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (placebo) (Placebo Comparator): Patients receive placebo oral solution (swish, gargle for 30 seconds, and slowly swallow) on day 1. Patients then crossover to Arm I on day 3.
  Interventions: Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Doxepin Hydrochloride — Given orally
  Other Names: Adapin; Sinequan
  Arms: Group I (doxepin hydrochloride)
Other: Placebo — Given orally
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies the effects of taking doxepin hydrochloride as compared to placebo (inactive drug) in treating esophageal pain in patients with cancer located in the chest area receiving radiation therapy to the thorax with or without chemotherapy. Doxepin hydrochloride is a tricyclic antidepressant drug which was recently shown to be helpful for mouth pain in patients receiving radiation therapy. Doxepin hydrochloride affects the surface of the esophagus, which may be helpful in reducing the pain caused by radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide baseline data regarding the effectiveness of doxepin (doxepin hydrochloride) in reducing esophagitis-related pain in patients undergoing radiation therapy (RT) to the thorax, as measured by a patient-reported questionnaire at 5 minutes, 15 minutes, 30 minutes, 1 hour and then at 2 and 4 hours on day 1.

SECONDARY OBJECTIVES:

I. To assess the adverse event profile of doxepin swish and swallow using a patient-reported questionnaire at 5 minutes, 15 minutes, 30 minutes, 1 hour and then at 2 and 4 hours using Common Terminology Criteria for Adverse Events (CTCAE) and Radiation Therapy Oncology Group (RTOG) acute toxicity criteria, and also for domains of unpleasant taste, burning/stinging discomfort, and drowsiness.

II. To evaluate the effectiveness of doxepin in reducing esophagitis-related pain in patients undergoing RT to the thorax, as measured by a patient-reported questionnaire at 5 minutes, 15 minutes, 30 minutes, 1 hours and then at 2 and 4 hours on days 1 and 3 (including the cross-over phase).

III. To compare and provide baseline data regarding alternative analgesic use between the doxepin and placebo arms.

IV. To provide baseline data regarding the patients? preference for continued therapy with doxepin or placebo after initial test dose or after the cross-over phase, as measured by items 9 and 10 in the patient-reported questionnaire at 4 hours after administration of the study medication and the actual participation rate.

TERTIARY OBJECTIVES:

I. To assess pain reduction and other adverse event profile in the optional continuation phase of doxepin oral rinse therapy. (Only applies to patients who have the optional continuation of doxepin oral rinse after the first two phases)

OUTLINE: Patients are randomized to 1 of 2 treatment groups.

GROUP I: Patients receive doxepin hydrochloride oral solution (swish, gargle for 30 seconds, and slowly swallow) on day 1. Patients then crossover to Arm II on day 3.

GROUP II: Patients receive placebo oral solution (swish, gargle for 30 seconds, and slowly swallow) on day 1. Patients then crossover to Arm I on day 3.

In both arms, patients may continue to receive doxepin hydrochloride oral solution every 4 hours as needed during radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of thoracic malignancies including non-small cell lung cancer (NSCLC), small lung cancer (SCLC), esophageal cancer, hypopharyngeal and laryngeal cancers (for which esophagitis symptoms can be relieved by doxepin swallow), lymphoma, thyroid, thymoma, thymic carcinoma, mesothelioma, sarcoma, and spinal, pulmonary or pleural-based metastases
* Planned RT (with or without chemotherapy) to a dose of >= 20 Gray (Gy) using 1.60 Gy per daily fraction; if radiation is given twice daily, a cumulative planned dose of >= 15 Gy using at least 1.25 Gy per fraction is required; hypofractionated and stereotactic body radiation therapy regimen are allowed
* At least 5 cm of the esophagus must be planned to receive radiotherapy, with a minimum dose of at least 10 Gy
* >= 3 esophageal pain, either at rest or during swallowing, felt to be related to esophagitis for which the patient wants relief, as measured by asking the following question

  * ?On a scale of 0 to 10 (0 = no pain; 10 = worst pain), what number best describes your chest pain* (right now) due to your radiation treatment??

    * Radiation can cause inflammation in your esophagus which can feel like a chest pain, either at rest or during swallowing
* Able to swallow the study medication
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Negative pregnancy test done =< 28 days prior to registration, for women of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willingness to complete evaluation and questionnaires per protocol at the participating institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Known allergy to doxepin, tricyclic antidepressants, or any known component of the drug formulation
* Histologic proof of and getting treatment for esophageal, stomach, spinal cord, thyroid, breast, and head and neck cancers and vertebral metastases
* Use of a tricyclic antidepressant or monoamine oxidase inhibitor within the 2 weeks prior to registration
* The presence or strong clinical suspicion of a tracheoesophageal fistula, or known esophageal invasion by cancer
* Current untreated or unresolved esophageal candidiasis or herpes simplex virus (HSV) infection
* Current untreated narrow angle glaucoma
* Current untreated urinary retention =< 6 weeks prior to registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Any of the following

  * Pregnant women
  * Nursing women
* Current use of doxepin or doxepin rinse as a swallow preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2017-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Sio, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 were accrued but only 3 provided data. Since only 1 patient was accrued & completed the study on 1 arm, patient confidentiality prevents the reporting of results per intervention. 2nd crossover was optional; none chose to crossover. The study results are only reported for the 1st study period (before crossover) & only for placebo intervention.
Groups:
- Placebo: Patients receive placebo oral solution (swish, gargle for 30 seconds, and slowly swallow) on day 1.
Period: Overall Study
Arm/Group | Placebo
Started | 3
Completed | 2
Not Completed | 1
Not completed — No treatment data | 1

BASELINE CHARACTERISTICS:
Population: 5 were accrued but only 3 provided data. Since only 1 patient was accrued & completed the study on 1 arm, patient confidentiality prevents the reporting of results per intervention. 2nd crossover was optional; none chose to crossover. The study results are only reported for the 1st study period (before crossover) & only for placebo intervention.
Arm/Group | Placebo
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 61.3 [53 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mouth Pain as Measured by Average Area Under the Curve Per Assessment
Description: Average Area Under the Curve per assessment (aAUCpa) of pain for the first cycle of treatment. Scores are reported on a 0-100 scale, where 100=better outcome QOL. The aAUCpa is the average of each AUC between each sequential assessment. Patients will assess their pain at baseline and at 5, 15, 30, 60, 120, and 240 minutes after treatment. The AUC calculation is based on the assessment number (1,2,3,4,5,6) instead of the actual number of minutes (5,15,30,60,120,240). This results in an AUC measure that is the average pain score across all of the measurements and is not a function of the number of minutes from treatment. The area under the curve of these 6 time points will be adjusted by their baseline pain score. The pain scores at each time point are given equal weights in the AUC calculation and the AUC calculation does not use the number of minutes after treatment. Therefore, the AUC measurement scale is the same as the original pain score scale.
Time Frame: Baseline and 5, 15, 30, 60, 120, and 240 minutes after treatment on day 1
Population: as for baseline characteristics
Measure: Number; unit: units on a scale
Arm/Group | Placebo
Number analyzed (Participants) | 3
units on a scale
  Patient #1 | -1.6
  Patient #2 | 0
  Patient #3 | NA — Patient did not report a baseline pain score, so an AUC adjusted for baseline could not be calculated.

2. Secondary Outcome: Incidence of Any Grade 3 or Higher Adverse Events Using Common Terminology Criteria for Adverse Events (CTCAE)
Description: Incidence of any grade 3 or higher adverse events using Common Terminology Criteria for Adverse Events (CTCAE). Number or patients reporting a grade 3 or higher adverse event according to CTCAE
Time Frame: Up to 4 hours after treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Use of Alternative Analgesics
Description: Subgroup analyses will be performed to determine differential effects within the two stratification factors.
Time Frame: Up to 4 hours after treatment
Population: Only patients who submitted data on alternative analgesics are evaluable for this outcome measure. None of the patients provided information about alternative analgesics, so this secondary outcome could not be analyzed.
Arm/Group | Placebo
Number analyzed (Participants) | 0

4. Secondary Outcome: Patient Preference for Continued Therapy at Initial Dose and Crossover
Time Frame: At initial Day 1 dose and Day 3 crossover dose.
Population: Only patients who submitted data on patient preference are evaluable for this outcome measure. Since none of the patients crossed over to the optional phase of the study, this secondary outcome could not be analyzed.
Arm/Group | Placebo
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Incidence of Adverse Events Graded According to Common Terminology Criteria for Adverse Events, Radiation Therapy Oncology Group, and Patient Reported Outcomes (Continuation Phase)
Description: Means and proportions, along with 95% confidence intervals and plots over time will be reported for adverse event levels by week.
Time Frame: Up to 3 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pain Levels (Continuation Phase)
Description: Means and proportions, along with 95% confidence intervals and plots over time will be reported for pain levels by week.
Time Frame: Up to 3 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Quality of Life Using European Organization for Research and Treatment of Cancer Quality of Life-Lung Cancer 13 and Functional Assessment of Cancer Therapy-Lung
Description: Comparative statistics will be used to explore the relationship between quality of life and radiation-induced thoracic toxicities. These analyses will include scatterplots, spearman correlations, t-tests and chi-square tests.
Time Frame: Up to 4 hours after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 hours after treatment on day 3
Description: Since only one patient was accrued and completed the study on one arm, patient confidentiality prevents the reporting of results per intervention. Therefore, the study results are only reported for the first study period (before crossover) and only for a single intervention (placebo).Serious AE (SAE) reports may include any serious or non-serious events considered related to the primary event; collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes